CLINICAL TRIAL: NCT05115981
Title: Psychoactive Drug Uses Among Medical and Pharmacy Students
Acronym: PSYCHO'ACT
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.161; 2020-A01352-37 (Other: ID RCB)
Record Dates: First submitted 2021-09-27; First posted 2021-11-10 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Psychoactive Substance Use Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Drug addiction to psychoactive substances, widely consumed in France, represents a major public health issue. The three main motivations identified for the consumption of psychostimulants would be self-medication, the party aspect and the improvement of school performance. Students of medicine and pharmacy are a population exposed to academic and professional stress, vulnerable to health problems and psycho-social disorders (anxiety, depression), with direct access to many drugs at their workplace. Almost a third of these students declared to consume these products to improve their cognitive performance, while a recent study showed that they take them instead to manage their stress and sleep. However, no study has characterized all the different uses of psychoactive drugs (PAD) in this population, nor the motivations for consumption, while an analysis of motives would help to develop better screening and prevention strategies. The main objective of the research is to characterize the motivations for PAD consumption among students of medicine and pharmacy in France. The most represented motives will be analyzed on the questionnaire of motivations for consumption (threshold frequency ≥20%). The secondary objectives are to identify the risk factors linked to the individual, to the environment and to drugs in students with PAD use disorders regardless of their motivation and in those using to improve their performance.

ELIGIBILITY:
Inclusion Criteria:

* Being of legal age
* Studying medicine or pharmacy in France from the 2nd to the 6th year
* Have read the newsletter and validated its no objection
* Have answered all the questions
* Validate the return of the questionnaire

Exclusion Criteria:

* partial filling of the online questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: medical and pharmacy students, from the 2nd to the 6th year, in France
Sampling Method: Non-Probability Sample
Enrollment: 1930 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
The main objective of the research is to characterize the motivations for psychoactive drugs consumption among medical and pharmacy students in France. | two months
  frequency of the most represented items concerning the main palatability drug on the Consumption Motivation Screening Questionnaire (frequency threshold considered ≥ 20%).
  (the minimum value of the questionnaire: 0 motivation of consumption; the maximum value: 110 motivations of consumption, higher scores mean a more severe addiction)

SECONDARY OUTCOMES:
In students with a psychoactive drug use disorder whatever their motivations, identify the risk factors related to the individual (anxiety) | two months
  assessment the intensity of anxiety on the Hospital Anxiety and Depression scale (the minimum value of the scale : 0 for Anxiety, 0 for Depression; the maximum value: 21 for Anxiety, 21 for depression; higher scores mean a worse outcome)
In students with a psychoactive drug use disorder whatever their motivations, identify the risk factors related to the individual (depression) | two months
  assessment the intensity of depression on the Hospital Anxiety and Depression scale (the minimum value of the scale : 0 for Anxiety, 0 for Depression; the maximum value: 21 for Anxiety, 21 for depression; higher scores mean a worse outcome)
In students with a psychoactive drug use disorder whatever their motivations, identify the risk factors related to the environment | two months
  family psychiatric history Psycho'act questionnaire
In students with a psychoactive drug use disorder whatever their motivations, identify the risk factors related to drugs. | two months
  assessment of the intensity of the psychoactive drug use disorder with the Addictive Intensity Evaluation Questionnaire (the minimum value of the questionnaire : 14; the maximum value: 98; higher scores mean a worse outcome)
In students with psychoactive drug use disorder for doping purposes, identify risk factors related to the individual (anxiety) | two months
  assessment the intensity of anxiety on the Hospital Anxiety and Depression scale (the minimum value of the scale : 0 for Anxiety, 0 for Depression; the maximum value: 21 for Anxiety, 21 for depression; higher scores mean a worse outcome)
In students with psychoactive drug use disorder for doping purposes, identify risk factors related to the individual (depression) | two months
  assessment the intensity of depression on the Hospital Anxiety and Depression scale (the minimum value of the scale : 0 for Anxiety, 0 for Depression; the maximum value: 21 for Anxiety, 21 for depression; higher scores mean a worse outcome)
In students with psychoactive drug use disorder for doping purposes, identify risk factors related to the environment | two months
  family psychiatric history Psycho'act questionnaire
In students with psychoactive drug use disorder for doping purposes, identify risk factors related to drugs. | two months
  assessment of the intensity of the psychoactive drug use disorder with the Addictive Intensity Evaluation Questionnaire (the minimum value of the questionnaire : 14; the maximum value: 98; higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble_Alpes UniversityHospital, Grenoble, France